CLINICAL TRIAL: NCT01311414
Title: Effect of Cafedrine/Theodrenaline and Urapidil During Carotid Endarterectomy on Cerebral Oxygenation Measured by Near Infrared Spectroscopy
Brief Title: Effect of Cafedrine/Theodrenaline and Urapidil on Cerebral Oxygenation
Acronym: NIRSMED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was suspended due to organizational problems
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Axel Fudickar, Dr. med., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudickar6
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Cerebral Ischemia
MeSH Terms: conditions — Brain Ischemia | interventions — cafedrine; theodrenaline; urapidil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cafedrine/theodrenalin (Experimental)
  Interventions: Drug: cafedrine/theodrenaline, urapidil

INTERVENTIONS:
Drug: cafedrine/theodrenaline, urapidil — Increasing blood pressure using cafedrine/theodrenalin and decreasing blood pressure using urapidil during carotid endarterectomy.

SUMMARY:
During clamping of one internal carotid artery for endarterectomy, blood flow through this vessel has to be compensated by collateral arteries including the contralateral internal artery and vertebral arteries. In 7 % of all patients undergoing carotid endarterectomy this collateral flow is not sufficient to maintain adequate cerebral perfusion during clamping and ischemic brain damage is likely to emerge. To maximize cerebral blood flow during clamping, increase of blood pressure is a common procedure and routine at our institution. Increasing blood pressure can be enabled by tapering a mixture of Cafedrine und Theodrenalin (Akrinor®) until the designated blood pressure is reached. After declamping, the blood pressure has to be reduced to normal values to avoid postoperative hyperperfusion syndrome. This is enabled by tapering urapidil until normal blood pressure is achieved.

It has been shown that cerebral oxygenation measured by near infrared spectroscopy is reduced by intravenous application of norepinephrine. Otherwise, intravenous nitroglycerine increases cerebral oxygenation during cardiopulmonary bypass. Hence, cafedrine/theodrenalin and urapidil may also have an effect on cerebral perfusion. In this prospective randomized study the effect of cafedrine/theodrenalin and urapidil on cerebral oxygenation measured by near infrared spectroscopy is investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for carotid endarterectomy

Exclusion Criteria:

* Cerebral disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygenation | 1 hour
  Outcome measure is change of cerebral oxygenation measured by near-infrared spectroscopy from values at baseline (arterial blood pressure in normal range) to values three minutes after increasing systolic blood pressure above 160 mmHg by intravenous injection of cafedrin/theodrenalin as needed (0,5 - 1 ml).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany